CLINICAL TRIAL: NCT06641375
Title: Anti-Reflux Endoscopic Therapy Using Argon Plasma Coagulation (AREA) in Gastroesophageal Reflux Disease (GERD) Patients
Brief Title: Anti-Reflux Endoscopic Therapy Using Argon Plasma Coagulation (AREA) in Gastroesophageal Reflux Disease (GERD) Patients: A Single Center, Randomized, Sham, Controlled Trial (The AREA Study)
Acronym: AREA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Mohan Ramchandani, STUDY DIRECTOR, Asian Institute of Gastroenterology, India
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AREA21
Record Dates: First submitted 2024-10-12; First posted 2024-10-15 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2024-10

CONDITIONS: GERD
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anti reflux endoscopic theraphy using Argon plasma coagulation in GERD (Active Comparator): To the intervention arm, the area of cardia, along greater curvature will be cleaned first followed by demarcation of a 1-1.5 cm area of non-ablation zone with two vertical lines by use of Pulsed APC using the H-APC catheter for marking and to prevent excess ablation . After this, the area of cardia, on either side will be injected in sequence using a combination of methylene blue and normal saline using the H-APC catheter jet system using between Effect 30 and Effect 70 on the ErbeJet 2 to raise the mucosa and create a submucosal cushion . Once adequate submucosal cushion is created, the mucosa starting below the z-line and up to 3 cm below will be treated by Pulsed APC 50W-80W using the H-APC catheter till golden-brown discoloration of the ablated tissue20
  The area of cardia below the Z-line will be treated in a 270-320-degree fashion. Once adequate ablation is achieved and no deeper tissue injury or bleeding is ensured, the procedure will be terminated.
  Interventions: Device: Anti reflux endoscopic theraphy
- Endoscopy (Placebo Comparator): Patients randomized to the control arm, will undergo a sham intervention. This will include performing upper endoscopy with procedural sedation followed by markings of landmarks as described. This will be followed by gastroscope retroflexion in the gastric cardia with at least 15 minute of examination time spent in retroflexion to reciprocate the H-APC intervention. No H-APC or submucosal injection or other intervention will be performed during the upper endoscopy with sham intervention. All Patients will also continue their PPI daily for 4 weeks.
  Interventions: Other: Endoscopy

INTERVENTIONS:
Device: Anti reflux endoscopic theraphy — o the intervention arm, the area of cardia, along greater curvature will be cleaned first followed by demarcation of a 1-1.5 cm area of non-ablation zone with two vertical lines by use of Pulsed APC using the H-APC catheter for marking and to prevent excess ablation . After this, the area of cardia, on either side will be injected in sequence using a combination of methylene blue and normal saline using the H-APC catheter jet system using between Effect 30 and Effect 70 on the ErbeJet 2 to raise the mucosa and create a submucosal cushion . Once adequate submucosal cushion is created, the mucosa starting below the z-line and up to 3 cm below will be treated by Pulsed APC 50W-80W using the H-APC catheter till golden-brown discoloration of the ablated tissue20
  The area of cardia below the Z-line will be treated in a 270-320-degree fashion. Once adequate ablation is achieved and no deeper tissue injury or bleeding is ensured, the procedure will be terminated.
  Arms: Anti reflux endoscopic theraphy using Argon plasma coagulation in GERD
Other: Endoscopy — Patients randomized to the control arm, will undergo a sham intervention. This will include performing upper endoscopy with procedural sedation followed by markings of landmarks as described. This will be followed by gastroscope retroflexion in the gastric cardia with at least 15 minute of examination time spent in retroflexion to reciprocate the H-APC intervention. No H-APC or submucosal injection or other intervention will be performed during the upper endoscopy with sham intervention. All Patients will also continue their PPI daily for 4 weeks.
  Arms: Endoscopy

SUMMARY:
Background and Rationale:

Gastroesophageal reflux disease is affecting 1 in 3 US adults with half experiencing daily symptoms. Per recent data, more than 50% continue to experience daily symptoms despite taking medical therapy and not eligible for surgery. In that small fraction of patients who are eligible for surgery, more than 70% resume taking a medicine for their reflux disease. GERD is common among the US veterans and currently there is a lack of minimally invasive endoscopic therapies for management of GERD. This study will investigate performance of minimally invasive, endoscopic therapy using antireflux mucosal ablation (hybrid argon plasma coagulation) that has been used in other areas of GI tract with efficacy and safety for management of chronic GERD among the US veterans.

Objective:

The aim of this study is to assess the safety and effectiveness of antireflux mucosal ablation or ARAT (intervention group) in patients with chronic gastroesophageal reflux disease (GERD) symptoms (typical symptoms of GERD, i.e. heartburn or acid reflux/regurgitation at least twice a week) for the last 6 months and objective evidence of reflux disease (positive ambulatory pH study off PPI for 5-7 days) compared to sham procedure (control group).

DETAILED DESCRIPTION:
Inclusion/Exclusion criteria: Inclusion:

* Patients with chronic GERD symptoms (at least 1 typical symptom of GERD, i.e. heartburn or acid reflux/regurgitation at least twice a week) for last 6 months and
* Objective evidence of reflux disease (positive ambulatory pH study)
* Patients prescribed standard dose of PPI for symptoms of GERD
* Able to undergo upper endoscopy as evidenced by completion of pre-endoscopy standard of care checklist.

Exclusion:

1. Patients unable to or unwilling to participate or consent
2. Age <18 years or >80 years
3. Allergic or intolerant to PPI medications
4. Large hiatal hernia > 3 cm and Hill grade IV
5. Barrett's esophagus
6. Esophageal stricture with any prior intervention
7. Major motility disorder on HRM

7. Eosinophilic esophagitis 8. Gastroparesis documented by abnormal gastric emptying time 9. Previous fundoplication, myotomy or LINX surgery 10. Cirrhosis with esophageal and/or gastric varices

Study groups:

Patients recruited will be randomized to undergo antireflux mucosal ablation (ARAT) OR sham intervention after inclusion and exclusion criteria have been met.

Study procedure:

Patients will be randomized (1:1) to one of the arms by computer generated random sequence of numbers.

The following study visits are foreseen for each patient:

Screening Visit(s) A screening visit is performed at the investigational site. During this visit out-patients will be informed about the aims, procedures, benefits and possible risks of the study prior to signing the informed consent form for inclusion in the study. Their medical history will be recorded as well as eventual clinical or laboratory examinations according to the local standard of care preparation for an upper endoscopy.

Randomization (Intervention) visit: Each eligible patient returns to the clinic to undergo either the study intervention OR sham intervention.

24-48 hour and 7-10 day post randomization phone call for adverse events among both groups.

25-30 day post randomization phone call for adverse events among both groups.

3-4 Month (80-112 days post randomization) visit with upper endoscopy and ambulatory pH monitoring to include administration of the validated GERD-HRQL and RDQ questionnaires

6-7 month (165-196 days post randomization) visit phone call to include administration of the validated GERD-HRQL and RDQ questionnaires

11-12 month (336-365 days post randomization) visit with upper endoscopy and ambulatory pH monitoring to include administration of the validated GERD-HRQL and RDQ questionnaires

1. To determine if ARAT can improve GERD-HRQL score 50% compared to sham intervention at 3, 6 and 12 months
2. To determine if ARAT can decrease GERD scores (RDQ) 50% compared to sham intervention at 3, 6 and 12 months

Secondary aims:

1. To determine if ARAT can reduce esophageal acid exposure time <4% (using wireless ambulatory 24-hr pH monitoring) in 50% subjects compared to sham intervention at 3 and 12 months
2. To determine if ARAT can achieve 50% reduction in DeMeester score compared to sham intervention at 3 and 12 months
3. To determine if ARAT can achieve PPI dose reduction or discontinuation in 25% of subjects after 3 months compared to sham intervention
4. To evaluate the safety profile of ARAT the rapy by recording major (GI bleeding, perforation, hospitalization, esophageal stricture) and minor complications (chest pain, fever, dysphagia) 7.5. Follow up Following the baseline assessment and performance of the upper endoscopy (either true intervention or sham), patients in both groups will be asked to complete the GERD-HRQL and RDQ questionnaires at 3 month ,6 month and 12 months using appropriate case report forms. In addition, the study staff will contact the patients by phone call at day 24- 48 hours, by phone call at 7-10 days and 25-30 days post procedure to record any adverse events. This will be accomplished using designated case report forms. At months 3 and 12, all patients will also undergo an upper endoscopy with assessment for

erosive esophagitis, and placement of pH capsule. During the 3 month, 6 month and 12 months visit, use of PPI therapy (dose and frequency) will be recorded. Response to therapy will be assessed using the following parameters: improvement of GERD-HRQL scores, reduction in RDQ scores, AET <4% and DeMeester score <14 (off PPI). Any patients with dysphagia after the ARAT will undergo repeat endoscopy for evaluation. If significant stricture, endoscopic dilation will be performed per severity of symptoms and stenosis.

Duration of this study from subject randomization to completion is 1 year, however, we anticipate study duration of at least 24 months for subject screening, completion of study visits and data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic GERD symptoms (at least 1 typical symptom of GERD, i.e. heartburn or acid reflux/regurgitation at least twice a week) for last 6 months and
* Objective evidence of reflux disease (positive ambulatory pH study)
* Patients prescribed standard dose of PPI for symptoms of GERD
* Able to undergo upper endoscopy as evidenced by completion of pre-endoscopy standard of care checklist.

Exclusion Criteria:

1. Patients unable to or unwilling to participate or consent
2. Age <18 years or >80 years
3. Allergic or intolerant to PPI medications
4. Large hiatal hernia > 3 cm and Hill grade IV
5. Barrett's esophagus
6. Esophageal stricture with any prior intervention
7. Major motility disorder on HRM

7. Eosinophilic esophagitis 8. Gastroparesis documented by abnormal gastric emptying time 9. Previous fundoplication, myotomy or LINX surgery 10. Cirrhosis with esophageal and/or gastric varices

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-02-10 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
AREA | 1 year
  To determine if procedure can decrease Gastroesophageal reflux scores (RDQ) 50% compared to sham intervention at 3, 6 and 12 months

SECONDARY OUTCOMES:
Anti reflux ablation theraphy | 365 days
  To determine if ARAT can achieve 50% reduction in DeMeester score compared to sham intervention at 3 and 12 months
AREA | 1 year
  To determine if ARAT can achieve PPI dose reduction or discontinuation in 25% of subjects after 3 months compared to sham intervention
Anti reflux ablation theraphy | 1 year
  To determine if intervention can reduce esophageal acid exposure time <4% (using wireless ambulatory 24-hr pH monitoring) in 50% subjects compared to sham intervention at 3 and 12 months
Reflux disease | 1 year
  To evaluate the safety profile of ARAT therapy by recording major (GI bleeding, perforation, hospitalization, esophageal stricture) and minor complications (chest pain, fever, dysphagia)

CONTACTS AND LOCATIONS:
Overall Officials: Mohan Dr Ramchandani, MBBS MD, Principal Investigator — Asian institute of Gastroenterology/AIG Hospitals; Kriti Dr Krishna, MBBS MD, Principal Investigator — AIG Hospitals
Locations (1):
- Asian Institute of Gastroenterology Hospital, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No